CLINICAL TRIAL: NCT00772564
Title: The Use of Statins for Myocardial Death Prevention: From Cell to Bedside
Brief Title: The Use of Statins for Myocardial Death Prevention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, N_Krivoy, Clinical Pharmacology Unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ator2685Hdm2[2]
Record Dates: First submitted 2008-10-11; First posted 2008-10-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Myocardial Infarction
Keywords: Acute ST Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 80 mg (Experimental)
  Interventions: Drug: Atorvastatin
- Atorvastatin 10 mg (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Oral Atorvastatin

SUMMARY:
The administration of high dose HMG-CoA reductase inhibitors (Statins) to patients with acute ST-elevation MI (hypoxia/ischemia) who are treated with primary PCI (reoxygenation/ reperfusion) will protect their cardiomyocytes from death and thus preserve LV ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from acute ST elevation resulting from myocardial infarction, Killip Classification 1 and 2 will be included at-random to either group. Included subjects should be able to give their informed consent to participate in this study.

Exclusion Criteria:

1. The impossibility to give the required informed consent.
2. Known allergy to Atorvastatin.
3. Base line serum creatinine of 1.4 mg/dL.
4. Killip Classification 3 and 4.
5. Persisting vomiting.
6. History of previous liver disease.
7. History of previous muscle disease or rabdomyolisis.
8. Treated already with high dose atorvastatin
9. Non Compliance.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Heart EcoCardiography and specific laboratory tests | Base line, second day and 60 days after myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Sammer Diab, MD, PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Haifa District, Israel